CLINICAL TRIAL: NCT04076163
Title: About the Efficacy of a Serious Game in Critical Appraisal Learning
Brief Title: About the Efficacy of a Serious Game in Critical Appraisal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mona mlika (Other)
Responsible Party: Sponsor-Investigator, mona mlika, Principal investigator, University Tunis El Manar
Organization: University Tunis El Manar (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1234
Record Dates: First submitted 2019-08-16; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Healthy Students

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): group of students participating to a face-to-face learning
- intervention group (Other): group of students using serious game
  Interventions: Other: serious game

INTERVENTIONS:
Other: serious game — a serious game was performed by the investigators in order to enhance the critical appraisal practice of students
  Arms: intervention group

SUMMARY:
Background: serious games have been reported as valuable method of learning since a decade. Even if their evident efficiency hasn't been always reported, their influence on the learners' motivation has become consensual. The authors aim to assess the efficacy of using serious games to teach critical appraisal practice to medical students in comparison to face-to-face learning methods.

Material and methods: the authors will perform a cluster randomised controlled trial including third-year medical students. Both groups will receive the same initial learning about elementary principals of evidence-based-medicine. Then, the control group will perform a critical appraisal of a case report and a recommendation article guided by a checklist and the intervention group performed a critical appraisal of the same manuscripts using a home-made serious game. Both groups will be invited to fulfil a multiple-choice-question test and a satisfaction likert-scale questionnaire.

DETAILED DESCRIPTION:
* Population: since 2013, 25 students in the third year of medical training are received in the Department of Pathology every year. The students were divided into 7 groups of 4 to 5 students with an interval period of 2 to 3 weeks between the different groups. The students were assigned randomly by the faculty of medicine of Tunis. The training period lasts three weeks according to the university's recommendations. All the students that were assigned by the faculty and who gave their consent to participate to this study were included. The students that were performing their training period in other Departments were excluded.
* Type of study: this is a cluster randomised controlled trial. This kind of randomization will be used because of the university board's assignment. It seems more comfortable to the tutor to use the same method of learning to every group.
* Intervention: this interventional and longitudinal study will be performed during a year-period. The students' groups will be randomly assigned to two groups by using computerised random number allocation and will be given the same pre and post test to answer. The test consists in a 7 general multiple-choice-questions in addition to 5 multi-choice questions related to a manuscript. Besides, The trainees will fulfil a Likert-type-scale satisfaction questionnaire to report their self-assessed competences and their motivation. Every suggestion will be coted between 1 to 4.
* Learning activities: training objectives are listed in the students' university portfolio. These objectives were performed by the faculty staff and validated by the pedagogical committee. The objectives were divided into items related to technical skills, the resolution of problems, ethical attitude and the critical appraisal of a scientific publication.

A diary about the daily activities of the students is available in the e-portfolio of the students. It contains their repartition in the Department and the different learning activities. Different methods of learning are displayed in the Department of Pathology including traditional methods which consisted in lectures dealing with the pathologies mentioned in the training board, integrative and participative methods consisting in case-based and problem-based learning.

The five steps of the evidence-based-practice (EBP) are planned during the third week. During the 4 initial days, the tutor will initiate the students to the elementary principles of evidence-based-medicine practice. Learning methods are mainly lecture-based. During the fifth day, groups that are randomized to the control group will participate to a workshop, which consisted in a collective critical appraisal session. The students will perform a critical appraisal of a case report and guidelines entitled: "Spontaneous regression of locally advanced non small cell lung cancer" and "Early and locally advanced non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up" (7,8). The choice of case report and recommendations was motivated by the fact that the students have never been practicing critical appraisal. The students will be given a checklist of the Tunisia medical journal (http://www.latunisiemedicale.com/) in order to facilitate this practice.

The intervention group will practice a critical appraisal of the same manuscript using the serious game developed by the tutor.

* Serious game: the authors developed a simulation-based serious game with design elements consisting in avatars, scores and explanations. This game was performed using itystudio software. The different scenes took place into a medical consultation. The students (players) have to choose the doctor's avatar. A realistic scenario was performed in order to include the approach of critical appraisal into a realistic health problem. The scenario performed was a 50-year-old-patient visiting his family doctor to explore an episode of haemoptysis. This episode was explored and the medical doctor had to announce the diagnosis of lung cancer to his patient. In order to explain the disease to the patient and to prepare him to the future investigations and to the treatment modalities, the doctor had to deal with a case report about a spontaneous regression of a lung cancer then recommendations of the ESMO. With every article downloaded by the students, a series of questions were asked and scored. When the students gave the good answers, the game continued and if they failed the game was over. Every student had the opportunity to repeat the game. Three competences were evaluated: announcing bad news, the critical appraisal of a case report and the critical appraisal of recommendations. Every competency was scored and the player received the final scores represented into 3 axes in the end of the game. The scenario established to perform the game is represented in figure 2. Some illustrations of the game are represented in figure 3. The game was also made available through the Department site link: https://sites.google.com/a/fmt.utm.tn/externes-services-d-anatomie-pathologique-prof-mezni/. The major characteristics of the game are represented in table 2.
* Statistics: statistical tests used to compare the scores between both groups consisted in student test with alpha levels set at 0.05. The authors used SPSS software (version 20.0).

ELIGIBILITY:
Inclusion Criteria:

* Third-year medical students
* Students in the department of Pathology

Exclusion Criteria:

* Other medical students
* Non consenting students

Ages: 20 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Critical appraisal score | 12 months
  10 multiple choice questions with score /20

SECONDARY OUTCOMES:
Satisfaction questionnaire | 12 months
  12 questions scaled from 1 to 4

CONTACTS AND LOCATIONS:
Locations (1):
- Mona Mlika, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No